CLINICAL TRIAL: NCT00486499
Title: I-125 Versus Pd-103 for Medium Risk Prostate Cancer
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: VA Puget Sound Health Care System (U.S. Federal Agency)
Collaborators: Dr. Gregory Merrick (Unknown); Theragenics Corporation (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 02-4407-V04
Record Dates: First submitted 2007-06-12; First posted 2007-06-14 (Estimated); Last update posted 2007-06-14 (Estimated); Status verified 2007-06

CONDITIONS: Prostate Cancer
Keywords: radiation; brachytherapy; prostate; cancer
MeSH Terms: conditions — Prostatic Neoplasms; Neoplasms

INTERVENTIONS:
Procedure: I-125 versus Pd-103 radioactive seed insertion

SUMMARY:
hypothesis: the shorter half-life of Pd-103 versus I-125, will increase the rate of tumor eradication.

A total of 660 patients with AJC clinical stage T1c-T2a prostatic carcinoma (Gleason grade 7 to 9 and/or PSA 10-20 ng/ml) will be randomized to implantation with I-125 (144 Gy) versus Pd-103 (124 Gy).

DETAILED DESCRIPTION:
Objective: The objective of this study is test the hypothesis that the shorter half-life of Pd-103 versus I-125, will increase the rate of tumor eradication.

Research plan:

A total of 660 patients with AJC clinical stage T1c-T2a prostatic carcinoma (Gleason grade 7 to 9 and/or PSA 10-20 ng/ml) will be randomized to implantation with I-125 (144 Gy) versus Pd-103 (124 Gy).

Methodology:

Randomization will be accomplished by the method of random permuted blocks.

Cancer status will be monitored by yearly serial serum PSA. Treatment-related morbidity will be monitored by personal interview, using standard American Urologic Association and Radiation Therapy Oncology Group criteria at 1, 3, 6, 12 and 24 months.

Primary endpoint: Time to treatment failure. Patients with serum PSA above 0.5 ng/ml two years or more after treatment will be considered to have residual or recurrent cancer and to have failed therapy.

ELIGIBILITY:
Inclusion Criteria:

* PSA 4-10 ng/ml
* Gleason score 5 or 6

Ages: 40 Years to 90 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 660 (Estimated)
Dates: Start 2003-03

PRIMARY OUTCOMES:
PSA-based cancer eradication

CONTACTS AND LOCATIONS:
Overall Officials: Kent E Wallner, MD, Principal Investigator — VA Puget Sound, Group Health Cooperative, U of Washington
Locations (2):
- United States (2):
  - Group Health Cooperative, Seattle, Washington
  - VA Puget Sound, Seattle, Washington